CLINICAL TRIAL: NCT04546464
Title: The Effects of Therapeutic Recreation Activities on Aberrant Behaviours of Individuals With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gaye Erkmen Hadi, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1234567
Record Dates: First submitted 2020-08-25; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Therapeutic Recreation; Intellectual Disability; Recreational Activities; Aberrant Behaviors
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Therapeutic Recreation Program (Experimental): The experimental recreation program, which consisted of two sessions per week and lasted approximately
  1 hour each session, lasted for 8 weeks between May 2019 and June 2019 for the adolescents in the experimental group. The Therapeutic Recreation Activity Program, which consists of 16 sessions, is organized according to the self-determination and entertainment development model. This model aims to provide individual development and prosperity by creating an entertaining environment with therapeutic recreation. According to the degree of enjoyment, activity improves freedom of choice, preferences and ability to express oneself. Pleasure is a feeling that the participant feels deeply during therapeutic recreation. Provides entertainment experience. Pleasure increases individual motivation to participate, as well as making the best use of physical, social and emotional conditions
  Interventions: Behavioral: Therapeutic Recreation Program
- Standard care (No Intervention)

INTERVENTIONS:
Behavioral: Therapeutic Recreation Program — The experimental recreation program, which consisted of two sessions per week and lasted approximately
  1 hour each session, lasted for 8 weeks between May 2019 and June 2019 for the adolescents in the experimental group. The Therapeutic Recreation Activity Program, which consists of 16 sessions, is organized according to the self-determination and entertainment development model. This model aims to provide individual development and prosperity by creating an entertaining environment with therapeutic recreation. According to the degree of enjoyment, activity improves freedom of choice, preferences and ability to express oneself. Pleasure is a feeling that the participant feels deeply during therapeutic recreation. Provides entertainment experience. Pleasure increases individual motivation to participate, as well as making the best use of physical, social and emotional conditions
  Arms: Experimental Therapeutic Recreation Program

SUMMARY:
The aim of this study was to determine the effect of Therapeutic Recreation Activities on Aberrant Behavior of Adolescents With Intellectual Disabilities.

The research was carried out at Meram Melike Hatun Special Education Vocational School in Konya. The study took place between May 2019 and June 2019. The parents of the participants who participated in the study consisted of the experimental group (n = 16) and the remaining parents (n = 16) formed the control group and the sample group (n = 32). The personal information form which measures demographic characteristics developed by the researchers according to the literature, and The Aberrant Behavior Checklist Scale were used. Data were analyzed in SPSS statistics 23 program. According to Shapiro Wilk test, sample group was not normal. For this reason, non-parametric tests were performed. In descriptive data, the mean, number, percentage will be used; Comparative statistics were made according to the assumptions of non-parametric test (Wilcoxon test, Mann Whitney U test). Therapeutic Recreation Activities was applied as total of 16 sessions, consisting of two sessions per week and each session lasting about 1 hour. The program was implemented by researcher.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Having a physical disability, Having Down syndrome

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The Aberrant Behavior Checklist total score | through study completion, an average of 1 year
  The Aberrant Behavior Checklist measures assessing treatment effects on maladaptive behaviors of the people with mental retardation
The sub-factor score level of the Aberrant Behavior Checklist have been labeled as follows: Hyperactivity. | through study completion, an average of 1 year
  Irritability, Agitation, Crying
The sub-factor score level of the Aberrant Behavior Checklist have been labeled as follows: Lethargy | through study completion, an average of 1 year
  Social Withdrawal
The sub-factor score level of the Aberrant Behavior Checklist have been labeled as follows: Stereotypic Behavior | through study completion, an average of 1 year
  repetitive or ritualistic movement, posture, or utterance.
The sub-factor score level of the Aberrant Behavior Checklist have been labeled as follows: Self-injury | through study completion, an average of 1 year
  self injurious behaviors
The sub-factor score level of the Aberrant Behavior Checklist have been labeled as follows: Others behaviors | through study completion, an average of 1 year
  The factor includes the following questions:
  Their requests must be fulfilled immediately. They have repeated conversations. His mood changes quickly. Likes to be apart from others

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Zengin, pHD, Study Chair — Researcher
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided